CLINICAL TRIAL: NCT02025751
Title: Phase 3 Companion Study of Intranasal Metoclopramide in Men With Symptomatic Diabetic Gastroparesis
Brief Title: Multicenter Study to Evaluate the Efficacy and Safety of Metoclopramide Nasal Spray in Men With Diabetic Gastroparesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evoke Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METO-IN-004
Record Dates: First submitted 2013-12-29; First posted 2014-01-01 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Gastroparesis
Keywords: Diabetes; Gastroparesis; Delayed gastric emptying; Nausea; Vomiting; Bloating; Abdominal pain; Early Satiety; Gastric stasis; Gastropathy
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis; Nausea; Vomiting; Abdominal Pain; Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoclopramide Nasal Spray (Experimental): Metoclopramide Nasal Spray 10 mg, 30 minutes before meals and at bedtime (QID) for 4 weeks
  Interventions: Drug: Metoclopramide Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): Placebo Nasal Spray 30 minutes before meals and at bedtime (QID) for 4 weeks
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Metoclopramide Nasal Spray — One 10 mg spray dose 30 minutes before meals and before bed for 28 days (QID)
  Arms: Metoclopramide Nasal Spray
Drug: Placebo Nasal Spray — One placebo spray dose 30 minutes before meals and before bed for 28 days (QID)
  Other Names: Vehicle
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is evaluate the safety and efficacy of Metoclopramide Nasal Spray compared to placebo in reducing the symptoms of diabetic gastroparesis in adult men.

DETAILED DESCRIPTION:
Diabetic men with clinical symptoms attributed to diabetic gastroparesis and documentation of delayed gastric emptying who meet the protocol-specified entry criteria will be randomized to Metoclopramide Nasal Spray 10 mg or placebo administered as a single intranasal spray four (4) times daily; 30 minutes before meals and at bedtime for a total of four (4) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 18 and 75 years
* Willingness and ability to give written informed consent
* The ability to read, understand and speak English
* Prior diagnosis of Type 1 or Type 2 diabetes
* Diagnosis of diabetic gastroparesis with confirmation of delayed gastric emptying
* A mean daily gastroparesis symptom score of ≥1.4 and ≤3.5 prior to randomization
* Willingness to discontinue current treatment for diabetic gastroparesis and to avoid all proscribed (excluded) medications, as specified by the protocol, for the duration of the study

Exclusion Criteria:

* Gastric bypass, gastric banding, gastric pacemaker, post surgical causes of gastroparesis and disorders known to be associated with abnormal gastrointestinal motility
* A history of allergic or adverse responses, including, but not limited to, acute dystonic reactions and tardive dyskinesia, to metoclopramide or any comparable or similar product
* A history of, or physical findings suggestive of, tardive dyskinesia
* A history of epilepsy or currently using and unwilling or unable stop other drugs known to be associated with extrapyramidal reactions at screening
* Malignancy (with the exception of treated squamous cell or basal cell carcinoma of the skin) currently present, initially diagnosed or recurring within five (5) years of screening
* Renal dysfunction calculated as creatinine clearance (CrCl) <40 mL/min at screening
* Hemoglobin A1c >11.5% at screening

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn R Carlson, DMD, MD, Study Director — Evoke Pharma, Inc.
Locations (49):
- United States (49):
  - Birmingham Gasteroenterology Associates, P.C., Birmingham, Alabama
  - Digestive Specialists of the Southeast, Dothan, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Central Arizone Medical Associates/Clinical Research Advantage, Mesa, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Precision Research Institute, LLC, Chula Vista, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Precision Research Institute, LLC, San Diego, California
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - International Research Associates, LLC, Miami, Florida
  - Advanced Medical Research, Port Orange, Florida
  - Tri-County Research, Athens, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Newton Medical Center, Conyers, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Indiana University Health UH 1634, Indianapolis, Indiana
  - Professional Research Network of Kansas, Wichita, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Kansas City Gastroenterology & Hepatology, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Premier Medical Group of the Hudson, PC, Poughkeepsie, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - LeBauer Research Associates, Greensboro, North Carolina
  - Kinston Medical Specialist Clinical Research Office, Kinston, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Dayton Gastroenterology, Beavercreek, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Lovelace Scientific Resources, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Burke Internal Medicine, Burke, Virginia
  - Manassas Clinical Research, Manassas, Virginia
  - National Clinical Research, Norfolk, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide Nasal Spray | Placebo Nasal Spray
Started | 26 | 27
Completed | 25 | 24
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 27 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53
Gastroparesis Symptom Assessment [Mean (Standard Deviation); unit: units on a scale] — Daily symptom diary collected using IVR
  units on a scale | 2.096 (0.4801) | 2.235 (0.4097) | 2.167 (0.4468)

OUTCOME MEASURES:

1. Primary Outcome: Gastroparesis Symptom Assessment (GSA), a Patient Reported Outcome Measure
Description: Change from the Baseline Period to Week 4 of the Treatment Period in the mean daily Gastroparesis Symptom Assessment (GSA) total score for subjects receiving Metoclopramide Nasal Spray 10 mg versus subjects receiving placebo. The GSA minimum value is 0 (no symptoms) and the maximum value is 4 (very severe symptoms). A higher score is a worse outcome.
Time Frame: Change from the Baseline Period to Week 4 in Daily Total Score (Intent-to Treat Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metoclopramide Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 26 | 27
score on a scale | -0.751 (0.4673) | -0.657 (0.9042)
Statistical Analysis 1: Comparison: Metoclopramide Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.597, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Metoclopramide Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 3/27
Other Adverse Events (participants affected / at risk) | 7/26 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide Nasal Spray (N=26) | Placebo Nasal Spray (N=27)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) — Worsening of gastroparesis
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Uncontrolled diabetes mellitus
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) — Abscess left shin (MRSA)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide Nasal Spray (N=26) | Placebo Nasal Spray (N=27)
Liver palpable (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study failed to meet recruitment goals (N=150) and was completed after 24 months (N=53). All study visits and assessments were completed. Limited pharmacokinetic (PK) samples so no calculated PK parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No